CLINICAL TRIAL: NCT05588947
Title: The Tele-Taking Charge After Stroke (TeleTaCAS) Randomized Controlled Feasibility Trial of Telehealth Take Charge vs Control
Brief Title: The Tele-Taking Charge After Stroke Randomized Controlled Feasibility Trial
Acronym: TeleTaCAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Sean Dukelow, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1.0 25Sept2022
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Stroke/Brain Attack
Keywords: self-determination; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Open Blinded Endpoint Feasibility Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-TaCAS (Experimental): Two Take Charge sessions delivered by telehealth six weeks apart, the first being at 2 to 16 weeks after stroke, the earliest possible time after discharge to the community.
  Interventions: Other: Take Charge session
- Control (Active Comparator): Life After Stroke: Survivor Stories video played by telehealth at 2 to 16 weeks after stroke, the earliest possible time after discharge to the community.
  Interventions: Other: Active Control

INTERVENTIONS:
Other: Take Charge session — A 'talk therapy' session designed to harness the person's self-determination, re-establishing purpose, identity, autonomy, and skills to Take Charge of their recovery after stroke
  Arms: Tele-TaCAS
Other: Active Control — Life After Stroke educational video
  Arms: Control

SUMMARY:
Take Charge is a novel, community-based treatment for stroke developed to harness a person's self-determination. Two prior clinical trials with 572 stroke survivors showed that Take Charge improves quality of life, independence, and social participation up to a year after stroke. Take Charge has also been shown to be overall cost-saving to the health system and is a useful adjunct to standard care after stroke.

Because of the COVID-19 pandemic, a lot of healthcare has moved into a telehealth approach. The simplicity of Take Charge may lend itself to being effective if delivered by telehealth, allowing greater access for people with stroke in rural communities. Improving the care we provide in underserved regions of the country is important to help the health of Canadians.

We are proposing a new study, working closely with the researchers who ran the previous Take Charge studies.

The goal of this feasibility clinical trial is to learn about Tele-Take Charge in adults with stroke who live in Southern Alberta. The main questions it aims to answer are:

* is delivering Take Charge by telehealth feasible?
* is Take Charge by telehealth acceptable to this population?

Participants will meet with facilitators online via Zoom at 4 to 16 weeks after stroke, and be randomized to receive either:

* two Tele-Take Charge sessions six weeks apart
* one control tele-education session.

Researchers will compare the Tele-Take Charge and control groups to see if there are any differences in outcome measures. these differences will help researchers to estimate the number of participants that will be needed for a larger, multi-centred effectiveness trial.

DETAILED DESCRIPTION:
For adults diagnosed with acute stroke who are discharged to community living (non-institutionalized), we wish to evaluate whether delivering two Take Charge sessions by telehealth is (1) acceptable to the population of Southern Alberta, and (2) feasible to do.

Subjects will be randomly assigned to receive either two Tele-Take Charge sessions or one tele-education session (Life After Stroke video) by telehealth (the active control).

The primary feasibility outcome will be recruitment rate. Secondary outcomes will be measured by a blinded outcomes assessor at 6 and 12 months, either by e-questionnaire or by telephone.

Those who received Tele-Take Charge will also be asked to complete an acceptability questionnaire, and will be invited to take part in an in-depth interview about their experience as part of a qualitative substudy.

ELIGIBILITY:
Inclusion Criteria:

* Discharged with diagnosis of stroke to non-institutionalised community living situation
* Answering 'No' to the question 'Are you fully recovered from your stroke?' (i.e., modified Rankin score [mRS] must be > 0)
* Able to access video calling with a smartphone, computer, or other device

Exclusion Criteria:

* Major comorbid illness that would dictate functional outcome at 12 months or life expectancy < 12 months
* Pre-stroke dependency (mRS > 2 before index stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | 12 months
  Number of participants recruited per month

SECONDARY OUTCOMES:
Eligibility | 12 months
  Number of people meeting eligibility criteria
Treatment adherence | 12 months
  Number receiving both sessions
Acceptability of Tele-TaCAS | 2 weeks after receiving Tele-TaCAS
  Participant acceptability questionnaire
Health-related quality of life | 6 and 12 months after stroke
  Physical Component Summary score of the Short Form 36
  The PCS of the SF-36 is a psychometrically robust measure of health-related quality of life. The score is formed from an algorithm comprising 36 questions that assess functional health and well-being from the perspective of the patient. The items contribute to eight health domains of physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. The eight domains all contribute to physical component summary (PCS) and mental component summary (MCS) scores. The minimal clinically important difference (MCID) of the PCS in stroke is estimated to be 2.5.
Independence - modified Rankin scale 0 to 2 | 6 and 12 months after stroke
  The modified Rankin scale (mRS) is a global disability measure used commonly in acute stroke trials. The scale ranges from 0 to 6. 0 = no symptoms, 1 = able to carry out all usual activities despite symptoms, 2 = able to look after own affairs without assistance but unable to carry out all usual activities, 3 moderate disability, unable to look after own affairs but able to walk without assistance, 4 = unable to attend to own bodily needs or unable to walk without assistance, 5 = severe disability, bedridden, 6 = dead.
Activities of Daily Living - Barthel Index | 6 and 12 months after stroke
  The Barthel Index (BI) measures a person's current ability to do 10 different common activities with or without assistance, including bathing, walking upstairs, toileting, and feeding. The total scores range from 0 to 20, with a higher score representing more independence.
Instrumental Activities of Daily Living / Social Participation - Frenchay Activities Index | 6 and 12 months after stroke
  The Frenchay Activities Index (FAI) is a measure of instrumental activities of daily living that assesses a broad range of activities associated with everyday life that a patient has participated in within the recent past. These can be separated into three domains: domestic chores, leisure/work, and outdoor activities. The patient self-reports how frequently each activity was done in the prior 3-6 months, and the total score can range from 0 to 45. The higher the score, the more social participation has been reported.
Quality of Life - EQ5D5L | 6 and 12 months after stroke
  European Quality of Life 5 Dimension 5 Levels (EQ-5D-5L) is a self-reported measure of global quality of life in five domains and at five levels. There is also a visual analogue scale from 0 - 100 to self-rate how healthy a person feels that particular day.
Self-Determination - AMP-C | 6 and 12 months after stroke
  An Autonomy Mastery Purpose Connectedness score derived by our group with four statements and self-reported level of agreement on a Likert scale. Not validated but measured in the last Take Charge trial.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Dr Vernon Fanning CareWest Rehabilitation Centre, Calgary
  - Foothills Medical Centre, Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Taking Charge After Stroke main results paper — https://pubmed.ncbi.nlm.nih.gov/32293236/